CLINICAL TRIAL: NCT01521195
Title: A Pilot Study of the Relationship Between Oxygen Delivery and Consumption During Extracorporeal Membrane Oxygenation.
Brief Title: Oxygen Consumption In Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000017147
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: pediatric; ECMO; extracorporeal blood flow; VO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients on veno-arterial (VA) ECMO (Experimental)
  Interventions: Device: Extracorporeal blood flow via ECMO machine

INTERVENTIONS:
Device: Extracorporeal blood flow via ECMO machine — Extracorporeal Membrane Oxygenation (ECMO) machine can provide complete support of heart and lung function.
  Extracorporeal blood flow will be given at baseline rate, increased by 25% and decreased by 25%

SUMMARY:
The investigators propose to examine the relationship between DO2 and VO2 in critically ill patients requiring an Extracorporeal Membrane Oxygenation (ECMO) machine. This machine can provide complete support of heart and lung function. In so doing, the investigators will be able to avoid physiologic coupling by increasing DO2 mechanically, by increasing blood flow through the ECMO circuit.

Null Hypothesis:

Increased oxygen delivery, by means of an increased rate of extracorporeal blood flow, is not associated with an increase in oxygen consumption.

Alternate Hypothesis:

Increased oxygen delivery, by means of an increased rate of extracorporeal blood flow, is associated with an increase in oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Critical Care Unit on veno-arterial ECMO.
* Hemodynamic stability established, as adjudged by the treating CCU staff physician.
* Informed consent by parent or legal guardian.
* Approval by treating CCU staff physician to approach parents/guardians for consent process at any given time.

Exclusion Criteria:

* Patients in the Critical Care Unit on veno-venous (VV) ECMO.
* Inability to tolerate study period without red cell transfusion.
* Presence of a large leak around the endotracheal tube (> 10% tidal volume).
* Patients requiring > 70 % FiO2 at the time of potential enrollment.
* Parent or legal guardian refuse consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | Baseline
  VO2 will be measured using a mass spectrometer as this is the gold standard.
Oxygen consumption (VO2) | 30min
  VO2 will be measured using a mass spectrometer as this is the gold standard.
Oxygen consumption (VO2) | 60min
  VO2 will be measured using a mass spectrometer as this is the gold standard.
Oxygen consumption (VO2) | 90min
  VO2 will be measured using a mass spectrometer as this is the gold standard.

SECONDARY OUTCOMES:
Arterial serum lactate level | Baseline, 30min, 60min, 90min
Oxygen extraction ratio. | Baseline, 30min, 60min, 90min

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kavanagh, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Tosoni A, La Rotta G, Breatnach C, Anand V, Foreman C, Davidson L, Redington AN, Kavanagh BP. Oxygen Delivery and Consumption Are Independent: Evidence from Venoarterial Extracorporeal Membrane Oxygenation in Resuscitated Children. Am J Respir Crit Care Med. 2015 Sep 15;192(6):765-7. doi: 10.1164/rccm.201502-0267LE. No abstract available. PMID 26371816